CLINICAL TRIAL: NCT01132066
Title: Pilot Study of Transcranial Direct Current Stimulation for Facilitating Swallowing Improvement After an Acute Unilateral Hemispheric Infarction
Brief Title: Transcranial Direct Current Stimulation (TDCS) for Facilitating Swallowing Improvement After an Acute Unilateral Hemispheric Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Sandeep Kumar, Assistant Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007P-000102
Record Dates: First submitted 2010-05-17; First posted 2010-05-27 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Dysphagia
Keywords: swallowing; stroke
MeSH Terms: conditions — Deglutition Disorders; Stroke | interventions — Transcranial Direct Current Stimulation; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tDCS (Experimental): tDCS will provide an increase in cortical excitability. Patients will be randomized to receive tDCS or sham stimulation.
  Interventions: Other: tDCS
- sham (Placebo Comparator): Sham stimulation will provide identical subjective sensation as anodal tDCS.
  Interventions: Other: Sham

INTERVENTIONS:
Other: tDCS — tDCS will lead to an increase in cortical excitability
  Arms: tDCS
Other: Sham — Sham will provide identical subjective sensation as tDCS
  Arms: sham

SUMMARY:
The purpose of the research study is to investigate the effect of a brain stimulation technique called Transcranial Direct Current Stimulation (TDCS) in improving swallowing functions in subjects who develop dysphagia after a unilateral hemispheric infarction.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* Between 24-168 hours after onset
* Moderate to severe dysphagia based on swallowing assessment

Exclusion Criteria:

* Preexisting swallowing impairment
* Intracerebral hemorrhage
* Pacemaker of other electrically sensitive device

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Dysphagia Outcome and Severity Scale Score (DOSS) | 5 days after study enrollment
  DOSS is a validated swallowing assessment scoring system that will rate the severity of dysphagia. It will be performed by a speech and swallow pathologist.

SECONDARY OUTCOMES:
Incidence of seizure | 5 days after study enrollment
  Number of patient having seizures during the 5 sessions of stimulation in either groups will be tabulated and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Kumar, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Kumar S, Wagner CW, Frayne C, Zhu L, Selim M, Feng W, Schlaug G. Noninvasive brain stimulation may improve stroke-related dysphagia: a pilot study. Stroke. 2011 Apr;42(4):1035-40. doi: 10.1161/STROKEAHA.110.602128. Epub 2011 Mar 24. PMID 21441148